CLINICAL TRIAL: NCT06584474
Title: THE EFFECT OF NEBULIZED AZITHROMYCIN AS AN ADJUVANT PREVENTIVE THERAPY FOR BRONCHOPULMONARY DYSPLASIA IN PRETERM INFANTS
Brief Title: THE EFFECT OF NEBULIZED AZITHROMYCIN AS THERAPY FOR BRONCHOPULMONARY DYSPLASIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Assistant professor of pediatrics at Alexandria University, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201867
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Bronchopulmonary Dysplasia; Premature; Ventilation, Mechanical
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I : Azithromycin group (Active Comparator): Patients will receive nebulized azithromycin (Xithrone, Amoun, Egypt) that will be initiated from day 7 of birth in a dose of 20 mg/kg/day in two divided doses for 3 weeks till the time of primary outcome assessment (at 28 days of age).
  Interventions: Drug: Azithromycin neubilization; Device: Lung ultrasound
- Group II: conventional treatment group (Placebo Comparator): Patients will not receive the medication, instead will receive 3 ml of nebulized normal saline as placebo control.
  Interventions: Device: Lung ultrasound

INTERVENTIONS:
Drug: Azithromycin neubilization — nebulized azithromycin (Xithrone, Amoun, Egypt) that will be initiated from day 7 of birth in a dose of 20 mg/kg/day in two divided doses for 3 weeks till the time of primary outcome assessment (at 28 days of age). Azithromycin solution for nebulization will be prepared from intravenous vials containing 500 mg lyophilized powder. First, each lyophilized powder vial will be prepared with 5 ml normal saline according to the manufacturer's instruction. The reconstituted solution will be diluted with 28.5 ml normal saline to make a final concentration of 17.5 mg/ml according to clinical pharmacy recommendation. For nebulization of azithromycin, 0.6 ml of final drug prepared solution will be taken for every
  1 kg body weight of patient, then made up to 3 ml of normal saline and will be administered by Aerogen Jet Nebulizer every 12 hours using 8 liter/min of medical air or by face mask if not mechanically ventilated. According to the manufacturer's declaration, prepared azithro
  Arms: Group I : Azithromycin group
Device: Lung ultrasound — Device A mobile device (PHILIPS ® HD11 XE) with a 10-MHz linear probe will be used for chest ultrasound. It will be done at day 14 of postnatal life.

SUMMARY:
The aim of the study is to determine the effectiveness of nebulized azithromycin therapy in prevention of BPD in very low birth weight preterm infants when compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age less than 32 weeks and birth weight less than 1500 g.
2. Infants who are still in need of respiratory support at day 7 of life (intubated, or by non-invasive mechanical ventilation, including CPAP and high-flow nasal cannula, or any form of oxygen therapy).

Exclusion Criteria:

* Gestational age ≥ 32 weeks.
* Newborns with congenital cyanotic heart diseases.
* Obvious major congenital malformations, known syndromes or chromosomal anomalies.
* Infants with signs compatible with the diagnosis of necrotizing enterocolitis (NEC) in the first week of life.
* Current use of steroids.

Ages: 7 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Development of BPD (bronchopulmonary dysplasia) | 28 days of life and/or 36 weeks postmenstrual age
  Developed BPD :Yes or No If patient fulfilled criteria of BPD ; patient is born at or less than 32 weeks gestational age and still need oxygen and or respiratory support at the 28 day or more postnatal age and/or 36 weeks postmenstrual age.
Lung Ultrasound assessment | 14 days postnatal age.
  Lung ultrasound score The score is calculated by the following points at different lung zones using lung ultrasound 0: A lines
  1. 3 or more nonconfluent B lines
  2. confluent B lines
  3. C profile or consolidation

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt